CLINICAL TRIAL: NCT01070576
Title: Arginine and Nitric Oxide (NO) Metabolism During Bone Healing and Non-union Development- Early Prognostic Markers
Brief Title: Arginine and Nitric Oxide (NO) Early Prognostic Markers for Non-union Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Martijn Poeze, MUMC+
Other Study IDs: MEC-09-2-123
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Fracture Healing; Atrophic Non Union Development; Hypertrophic Non Union Development
Keywords: non union; fracture; healing; arginine; NO
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone debris and bloodsamples for amino acid determination
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- normal fracture healing: group in which normal fracture healing has occured
  Interventions: Other: no intervention
- atrophic: patients in which an atrophic non-union occured
  Interventions: Other: no intervention
- hypertrophic: patients in which a hypertrophic non-union occured
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Objective: Primary objective is to study the arginine-NO metabolism during fracture healing and dysfunctional fracture healing. Secondary objective: to investigate if differences or decreased arginine and NO concentrations in bone healing form a prognostic marker for non-union development Hypothesis: Early detection of disturbances in the Arginine and nitric oxide metabolism during fracture healing are a good prognostic marker for non-union development.

Study design: Prospective observational study. Study population: All acute fracture patients (age >18 years), with a fracture of the tibia or femur attending the Department of General Surgery, to investigate the Arginine -NO metabolism during normal fracture healing and possible dysfunctional healing. In total 100 patients will be included during this study.

Main study parameters/endpoints:

Primary endpoints are arginine and Nitric Oxide levels in the plasma during normal and dysfunctional fracture healing the bone in patients with and without non-union Secondary endpoints are levels of Nitric Oxide citrulline, ornithine and other amino acids in bone and in plasma Other parameters: baseline demography details will be obtained, including possible confounders, such as bodyweight, smoking, alcohol abuse, which may interfere with the outcome of this study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The extent of the burden and risk associated with participation is expected to be low during this study. In total, 7 blood samples will be taken during this study (45ml, in total). During the primary (and possible secondary) surgical procedure, bone debris will be taken. Bone debris is usually discarded but will be used for analysis in this study. There is no extra surgical procedure necessary to obtain the bone debris.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Patient with a fracture of the femur or tibia for which a surgical procedure providing bone debris is performed as therapy

Exclusion Criteria:

* Patients with another bone fracture in their recent medical history
* Infectious complications, such as infected pseudo-arthrosis
* Use of chronic corticosteroids or nitrovasodilating medication
* Patients with severe metabolic disturbances (liver, and renal insufficiency, diabetes).
* Patients with metastases, haematological malignancies or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute fracture of the femur or tibia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The arginine, NO, citrulline and ornithine levels in plasma and bone debris during normal and dysfunctional fracture healing in patients with and without a non-union | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Poeze, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands